CLINICAL TRIAL: NCT00250081
Title: Multi Center Project: Comparison of Functional Outcomes of Tendon Transfer Surgery, Botulinum Toxin Injections and Regular Ongoing Treatment in Hemiplegic Upper Extremity Cerebral Palsy
Brief Title: Comparison of Tendon Transfer, Botox Injections and Ongoing Treatment in Hemiplegic Cerebral Palsy
Acronym: UECP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual is complete.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michelle James, Chief of Orthopaedics, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 83004-278826
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Tendon Transfer; Botulinum Toxin Type A; Occupational Therapy; Child
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Therapy Group (Active Comparator): Therapy only
  Interventions: Procedure: Regularly ongoing therapy
- Surgery Group (Active Comparator): surgical intervention
  Interventions: Procedure: Upper Extremity Tendon transfer
- Botox Injections (Active Comparator): botulinum toxin
  Interventions: Procedure: Botulinum Toxin injections in Upper Extremity

INTERVENTIONS:
Procedure: Upper Extremity Tendon transfer
  Arms: Surgery Group
Procedure: Botulinum Toxin injections in Upper Extremity
  Arms: Botox Injections
Procedure: Regularly ongoing therapy
  Arms: Therapy Group

SUMMARY:
Doctors use different treatments for people with Cerebral Palsy. Surgery is one option. Botulinum toxin injections are another option; these are given directly into spastic muscles to weaken them temporarily. Regular ongoing treatment (splinting, stretching and exercises) is another option. The investigators want to find out if surgery works better than Botulinum Toxin (Botox) injections or regular ongoing treatment (therapy), and if the effects of Botulinum Toxin injections last for longer than six months.

DETAILED DESCRIPTION:
The specific aims of this study and the methodology for achieving them are:

1. To determine if tendon surgery for the forearm, wrist and thumb deformities of UECP is more effective than Botulinum toxin injections or regular ongoing treatment at improving function and quality of life for children with UECP. Children who are candidates for tendon surgery will be prospectively randomized to one of three treatment groups: standard tendon surgery, a series of three Botulinum toxin injections over a period of 12 months, and regular ongoing treatment. Validated tests of cognition, function and quality of life with tests of stereognosis and range of motion will be administered before, during and after treatment in order to compare outcomes of the three treatment groups.
2. To determine if serial Botulinum toxin injections have long-term beneficial effects on upper extremity function which outlast their paralytic effects.

Botulinum toxin has been shown to have beneficial effects on UE function while the muscles injected remain weakened by the toxin. Clinicians have theorized that improvements in UE function are maintained after the toxin wears off, but this has not been proven. Children randomized to the Botulinum toxin injection group will receive 3 injections. Their function will be tested before the first injection, while the paralytic results of the second injection are still in effect, and after the paralytic effects of the third injection have worn off, and the results compared in order to determine if functional improvements outlast the medicinal effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of UECP
* aged four to 17 years
* candidate for standard surgical management (tendon transfer)

Exclusion Criteria:

* subject could benefit from procedures in addition to standard surgical management and releases, and these procedures could be performed at the same anesthetic (for example, elbow flexor release)
* previous Botulinum toxin injection session in the affected UE in < 1 year
* previous ipsilateral UE surgery
* primary language other than English or Spanish
* subject and/or parent unwilling to attend eight therapy sessions and perform home exercise protocol

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2005-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Shriners Hospitals Upper Extremity Evaluation (SHUEE) | Initial, 6 mon, 1 year
Box & Blocks | Initial, 6 mon, 1 year
Assisting Hand Assessment (AHA) | Initial, 6 mon, 1 year

SECONDARY OUTCOMES:
Scores on questionnaires that assess participation and patient satisfaction at initial, 6 month and 1 year post intervention. | Initial, 6 mon, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michelle James, MD, Principal Investigator — Shriners Hospitals for Children, Northern Calfiornia; Ann Van Heest, MD, Principal Investigator — Shriners Hospitals for Children, Twin Cities; Anita Bagley, PhD, Principal Investigator — Shriners Hospitals for Children, Northern California
Locations (10):
- United States (10):
  - Shriners Hospitals for Children Northern California, Sacramento, California
  - Alfred I duPont Childrens Hospital, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shriners Hosptials for Children, Tampa, Florida
  - Shriners Hospitals for Children Chicago, Chicago, Illinois
  - Shriners Hospitals for Children, Shreveport, Louisiana
  - Shriners Hospitals for Children, Twin Cities, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Shriners Hospitals for Children, Greenville, South Carolina
  - Shriners Hosptials for Children, Intermountain, Salt Lake City, Utah

REFERENCES:
- [Background] BAX MC. TERMINOLOGY AND CLASSIFICATION OF CEREBRAL PALSY. Dev Med Child Neurol. 1964 Jun;6:295-7. doi: 10.1111/j.1469-8749.1964.tb10791.x. No abstract available. PMID 14155190
- [Background] Autti-Ramo I, Larsen A, Taimo A, von Wendt L. Management of the upper limb with botulinum toxin type A in children with spastic type cerebral palsy and acquired brain injury: clinical implications. Eur J Neurol. 2001 Nov;8 Suppl 5:136-44. doi: 10.1046/j.1468-1331.2001.00046.x. PMID 11851742
- [Background] Autti-Ramo I, Larsen A, Peltonen J, Taimo A, von Wendt L. Botulinum toxin injection as an adjunct when planning hand surgery in children with spastic hemiplegia. Neuropediatrics. 2000 Feb;31(1):4-8. doi: 10.1055/s-2000-15289. PMID 10774988
- [Background] Wall SA, Chait LA, Temlett JA, Perkins B, Hillen G, Becker P. Botulinum A chemodenervation: a new modality in cerebral palsied hands. Br J Plast Surg. 1993 Dec;46(8):703-6. doi: 10.1016/0007-1226(93)90203-n. PMID 8298785
- [Background] Wallen MA, O'flaherty SJ, Waugh MC. Functional outcomes of intramuscular botulinum toxin type A in the upper limbs of children with cerebral palsy: a phase II trial. Arch Phys Med Rehabil. 2004 Feb;85(2):192-200. doi: 10.1016/j.apmr.2003.05.008. PMID 14966702
- [Background] Fehlings D, Rang M, Glazier J, Steele C. An evaluation of botulinum-A toxin injections to improve upper extremity function in children with hemiplegic cerebral palsy. J Pediatr. 2000 Sep;137(3):331-7. doi: 10.1067/mpd.2000.108393. PMID 10969256
- [Background] El-Said NS. Selective release of the flexor origin with transfer of flexor carpi ulnaris in cerebral palsy. J Bone Joint Surg Br. 2001 Mar;83(2):259-62. doi: 10.1302/0301-620x.83b2.10763. PMID 11284577
- [Background] Hoffer MM, Lehman M, Mitani M. Long-term follow-up on tendon transfers to the extensors of the wrist and fingers in patients with cerebral palsy. J Hand Surg Am. 1986 Nov;11(6):836-40. doi: 10.1016/s0363-5023(86)80232-5. PMID 3794239
- [Background] Thometz JG, Tachdjian M. Long-term follow-up of the flexor carpi ulnaris transfer in spastic hemiplegic children. J Pediatr Orthop. 1988 Jul-Aug;8(4):407-12. doi: 10.1097/01241398-198807000-00005. PMID 3392191
- [Background] Tonkin M, Gschwind C. Surgery for cerebral palsy: Part 2. Flexion deformity of the wrist and fingers. J Hand Surg Br. 1992 Aug;17(4):396-400. doi: 10.1016/s0266-7681(05)80261-x. PMID 1402265
- [Background] Wenner SM, Johnson KA. Transfer of the flexor carpi ulnaris to the radial wrist extensors in cerebral palsy. J Hand Surg Am. 1988 Mar;13(2):231-3. doi: 10.1016/s0363-5023(88)80055-8. PMID 3351249
- [Background] Wolf TM, Clinkscales CM, Hamlin C. Flexor carpi ulnaris tendon transfers in cerebral palsy. J Hand Surg Br. 1998 Jun;23(3):340-3. doi: 10.1016/s0266-7681(98)80054-5. PMID 9665522
- [Background] Beach WR, Strecker WB, Coe J, Manske PR, Schoenecker PL, Dailey L. Use of the Green transfer in treatment of patients with spastic cerebral palsy: 17-year experience. J Pediatr Orthop. 1991 Nov-Dec;11(6):731-6. doi: 10.1097/01241398-199111000-00006. PMID 1960196
- [Background] Strecker WB, Emanuel JP, Dailey L, Manske PR. Comparison of pronator tenotomy and pronator rerouting in children with spastic cerebral palsy. J Hand Surg Am. 1988 Jul;13(4):540-3. doi: 10.1016/s0363-5023(88)80091-1. PMID 3418056
- [Background] Manske PR. Redirection of extensor pollicis longus in the treatment of spastic thumb-in-palm deformity. J Hand Surg Am. 1985 Jul;10(4):553-60. doi: 10.1016/s0363-5023(85)80082-4. PMID 4020069
- [Background] Hoffer MM, Perry J, Melkonian G. Postoperative electromyographic function of tendon transfers in patients with cerebral palsy. Dev Med Child Neurol. 1990 Sep;32(9):789-91. doi: 10.1111/j.1469-8749.1990.tb08482.x. PMID 2227142
- [Background] Perry J, Hoffer MM. Preoperative and postoperative dynamic electromyography as an aid in planning tendon transfers in children with cerebral palsy. J Bone Joint Surg Am. 1977 Jun;59(4):531-7. PMID 863949
- [Background] Hoffer MM. The use of the pathokinesiology laboratory to select muscles for tendon transfers in the cerebral palsy hand. Clin Orthop Relat Res. 1993 Mar;(288):135-8. PMID 8458126
- [Background] Kozin SH, Keenan MA. Using dynamic electromyography to guide surgical treatment of the spastic upper extremity in the brain-injured patient. Clin Orthop Relat Res. 1993 Mar;(288):109-17. PMID 8458122
- [Background] Mowery CA, Gelberman RH, Rhoades CE. Upper extremity tendon transfers in cerebral palsy: electromyographic and functional analysis. J Pediatr Orthop. 1985 Jan-Feb;5(1):69-72. doi: 10.1097/01241398-198501000-00012. PMID 3980710
- [Background] Johanson ME, James MA, Skinner SR. Forearm muscle activation during power grip and release. J Hand Surg Am. 1998 Sep;23(5):938-44. doi: 10.1016/S0363-5023(98)80177-9. PMID 9763276
- [Background] Johanson ME, Skinner SR, Lamoreux LW. Phasic relationships of the intrinsic and extrinsic thumb musculature. Clin Orthop Relat Res. 1996 Jan;(322):120-30. PMID 8542687
- [Background] Johanson ME, Skinner SR, Lamoreux LW, St Helen R, Moran SA, Ashley RK. Phasic relationships of the extrinsic muscles of the normal hand. J Hand Surg Am. 1990 Jul;15(4):587-94. doi: 10.1016/s0363-5023(09)90020-x. PMID 2380522
- [Background] Palmieri TL, Petuskey K, Bagley A, Takashiba S, Greenhalgh DG, Rab GT. Alterations in functional movement after axillary burn scar contracture: a motion analysis study. J Burn Care Rehabil. 2003 Mar-Apr;24(2):104-8. doi: 10.1097/01.BCR.0000054170.62555.09. PMID 12626930
- [Background] Rab G, Petuskey K, Bagley A. A method for determination of upper extremity kinematics. Gait Posture. 2002 Apr;15(2):113-9. doi: 10.1016/s0966-6362(01)00155-2. PMID 11869904
- [Background] Mosqueda T, James MA, Petuskey K, Bagley A, Abdala E, Rab G. Kinematic assessment of the upper extremity in brachial plexus birth palsy. J Pediatr Orthop. 2004 Nov-Dec;24(6):695-9. doi: 10.1097/00004694-200411000-00018. PMID 15502572
- [Background] Albright AL, Barry MJ, Painter MJ, Shultz B. Infusion of intrathecal baclofen for generalized dystonia in cerebral palsy. J Neurosurg. 1998 Jan;88(1):73-6. doi: 10.3171/jns.1998.88.1.0073. PMID 9420075
- [Background] Fedrizzi E, Pagliano E, Andreucci E, Oleari G. Hand function in children with hemiplegic cerebral palsy: prospective follow-up and functional outcome in adolescence. Dev Med Child Neurol. 2003 Feb;45(2):85-91. PMID 12578233
- [Background] Law M, King G. Parent compliance with therapeutic interventions for children with cerebral palsy. Dev Med Child Neurol. 1993 Nov;35(11):983-90. doi: 10.1111/j.1469-8749.1993.tb11580.x. PMID 8224565
- [Background] Manske PR, Langewisch KR, Strecker WB, Albrecht MM. Anterior elbow release of spastic elbow flexion deformity in children with cerebral palsy. J Pediatr Orthop. 2001 Nov-Dec;21(6):772-7. PMID 11675553
- [Background] Rodriquez AA, McGinn M, Chappell R. Botulinum toxin injection of spastic finger flexors in hemiplegic patients. Am J Phys Med Rehabil. 2000 Jan-Feb;79(1):44-7. doi: 10.1097/00002060-200001000-00010. PMID 10678602
- [Background] Tonkin MA, Hatrick NC, Eckersley JR, Couzens G. Surgery for cerebral palsy part 3: classification and operative procedures for thumb deformity. J Hand Surg Br. 2001 Oct;26(5):465-70. doi: 10.1054/jhsb.2001.0601. PMID 11560430
- [Background] Van Heest AE, House JH, Cariello C. Upper extremity surgical treatment of cerebral palsy. J Hand Surg Am. 1999 Mar;24(2):323-30. doi: 10.1053/jhsu.1999.0323. PMID 10194018
- [Background] Bourke-Taylor H. Melbourne Assessment of Unilateral Upper Limb Function: construct validity and correlation with the Pediatric Evaluation of Disability Inventory. Dev Med Child Neurol. 2003 Feb;45(2):92-6. PMID 12578234
- See also: Official website for Shriners Hospitals for Children, a network of 22 hospitals that provide expert, no-cost orthopaedic and burn care to children under 18 — http://www.shrinershq.org/Hospitals/Main